CLINICAL TRIAL: NCT00062933
Title: A Phase II Study of Isolated Hepatic Perfusion (IHP) With Melphalan Followed by Temozolomide for Subjects With Unresectable Hepatic Metastases From Ocular Melanoma
Brief Title: A Phase II Study of Isolated Hepatic Perfusion (IHP) in Patients With Ocular Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030221; 03-C-0221; NCT00066521 (obsolete NCT alias)
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Melanoma
Keywords: Clinical Response; Duration of Response; Quality of Life; Hyperthermia; Survival; Melanoma; Ocular Melanoma; Eye Cancer
MeSH Terms: conditions — Melanoma; Hyperthermia; Uveal Melanoma; Eye Neoplasms | interventions — Laparotomy

INTERVENTIONS:
Procedure: Laparotomy

SUMMARY:
Ocular melanoma, or cancer of the eye, is a rare form of cancer that can spread to the liver. A tumor in the liver, because of its size or location, sometimes cannot be removed with surgery.

The purpose of this study is to determine whether chemotherapy delivered only to the liver, called isolated hepatic perfusion (IHP), followed by systemic (to the whole body) chemotherapy improves the ability to treat cancer.

Study participants must be 18 years or older and have ocular melanoma that has spread to the liver. Before enrolling in the study, they will undergo the following evaluations: a physical exam; x-rays; blood tests; electrocardiogram; computed tomography (CT) scan of the chest, abdomen and pelvis; and a magnetic resonance imaging (MRI) scan of the liver.

The study includes a 15-minute quality-of-life questionnaire. Participants will complete the questionnaire 7 times over a period of 2 years to help investigators gauge their health status and progress.

A laparotomy is done, which allows a surgeon to view the tumor in the liver through a small incision in the abdomen while the patient is under general anesthesia. Sometimes the tumor can spread outside the liver in a way that cannot be seen by pre-operative scans. When this happens, the participant is ineligible to continue in the study, since an important part of the treatment is given only to the liver.

If the laparotomy reveals that the participant is eligible for the remainder of the study, the participant will receive IHP treatment during the surgery. Plastic tubes called catheters are placed in the vein and artery that feed and drain the liver. This creates a separate blood supply for the liver alone. Heated chemotherapy is then given into the liver blood supply for one hour, while being carefully kept out of the rest of the body.

After recovering from the surgery, eligible participants will receive a systemic chemotherapy called temozolomide for up to one year. This chemotherapy is taken by mouth in capsule form.

Participants will be asked to return to NIH 10-11 times during the first year to evaluate their progress.

DETAILED DESCRIPTION:
Patients with unresectable hepatic metastases secondary to ocular melanoma will undergo a 60 minute hyperthermic isolated hepatic perfusion with 1.5mg/kg melphalan followed by up to one year of oral temozolomide. Response to treatment, duration of response, patterns of failure, survival, and quality of life end-points will be followed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Histologically or cytologically proven measurable metastatic ocular melanoma confined to the liver. Patients with limited sites of extra-hepatic disease and who have dominant life-limiting disease in liver will be considered eligible if the extra-hepatic sites can be treated with local ablative measures such as resection or external beam radiation therapy. Patients with limited extra-hepatic disease will undergo IHP and treatment of extra-hepatic disease in a sequence determined by the clinical presentation but all patients will have had all disease treated prior to initiating temozolomide therapy.

Patients must have had no chemotherapy, radiotherapy, or biologic therapy for their malignancy for 28 days prior to the liver perfusion and must have recovered from all side effects except those outlined in appendix III.

Patients must have an ECOG performance standard of 0,1 or 2 prior to on-study and on the day prior to treatment with IHP.

Patients must have adequate hepatic function as evidenced by bilirubin less than 2.0 mg/dL and a PT equal to 2 seconds of the upper normal limit AST/ALT less than or equal to 10 times ULN.

Patients must be 18 years of age or greater and must be greater than 30 kg, because of reason outlined in Section 6.2.

Patients must have a platelet count greater than 75,000, a HCT greater than 27.0, an ANC greater than or equal to 1,500/ul, and a creatinine less than or equal to 1.5 mg/dL unless the measured creatinine clearance is greater than 60 mL/min/1.73 m(2).

Patients must be aware of the neoplastic nature of his/her illness, the experimental nature of the therapy , alternative treatments, potential benefits, and risks. The patient must be willing to sign an informed consent.

EXCLUSION CRITERIA:

Pregnant patients and nursing mothers will be excluded due to the unknown effects of melphalan on the fetus or newborn.

Patients taking immunosuppressive drugs or on chronic anticoagulation will not be eligible.

Patients with active systemic infections are not eligible.

Patients with biopsy proven cirrhosis or evidence of significant portal hypertension by history, endoscopy, or radiologic studies will be excluded.

Patients with a history of congestive heart failure with an LVEF less than 40% will be excluded.

Patients with COPD or other chronic pulmonary disease with PFT's less than 50% predicted for age will be excluded.

Patients with a history or diagnosis of veno-occlusive disease (VOD) will be excluded.

Patients with chronic active hepatitis based on a positive serology test for surface antigen B or C will be excluded if there is evidence of cirrhosis on pathology. If no pathology specimen exists then evidence for cirrhosis will be determined based on radiological studies and physical examination. If there are no indications of it then the patient will be registered on study and a biopsy will be obtained at the time of laparotomy for IHP with the expectation that occult clinically significant cirrhosis is very unlikely. If cirrhosis is pathologically confirmed the patient will not undergo treastment and be taken off study. Patients with radiographic or other signs of cirrhosis will undergo percutaneous biopsy prior to registration.

Patients with a prior hypersensitivity reaction to melphalan, dacarbazine, or temozolomide will be ineligible for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Becker JC, Terheyden P, Kampgen E, Wagner S, Neumann C, Schadendorf D, Steinmann A, Wittenberg G, Lieb W, Brocker EB. Treatment of disseminated ocular melanoma with sequential fotemustine, interferon alpha, and interleukin 2. Br J Cancer. 2002 Oct 7;87(8):840-5. doi: 10.1038/sj.bjc.6600521. PMID 12373596
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2003-C-0221.html